CLINICAL TRIAL: NCT02314546
Title: Intranasal Midazolam in Children as a Pre-Operative Sedative
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, David A Ullman MD, Attending Physician - Anesthesiology, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 994
Record Dates: First submitted 2014-12-03; First posted 2014-12-11 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Sedation, Conscious
MeSH Terms: interventions — Midazolam; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline placebo (Placebo Comparator): saline placebo
  Interventions: Drug: saline placebo
- Nasal Midazolam only (Active Comparator): Nasal Midazolam only - Patients received 0.2 mg/kg of intranasal midazolam
  Interventions: Drug: Midazolam
- Midazolam and Xylocaine (Active Comparator): Midazolam Plus Xylocaine - Patients received 0.2 mg/kg intranasal midazolam plus xylocaine 4% in a dose based on 25% of the volume of the midazolam
  Interventions: Drug: Midazolam; Drug: xylocaine

INTERVENTIONS:
Drug: Midazolam — Study participants will be randomly assigned to one of three treatment groups:
  * Group 1 - Placebo - Control patients will receive intranasal saline.
  * Group 2 - Nasal Midazolam Only - Patients will receive 0.2 mg/kg of intranasal midazolam.
  * Group 3 - Midazolam Plus Xylocaine - Patients will receive 0.2 mg/kg intranasal midazolam plus xylocaine 4% in a dose based on 25% of the volume of the midazolam.
  Other Names: versed
  Arms: Midazolam and Xylocaine; Nasal Midazolam only
Drug: xylocaine — Midazolam Plus Xylocaine - Patients will receive 0.2 mg/kg intranasal midazolam plus xylocaine 4% in a dose based on 25% of the volume of the midazolam.
  Arms: Midazolam and Xylocaine
Drug: saline placebo — Placebo - Control patients will receive intranasal saline.
  Arms: Saline placebo

SUMMARY:
The purpose of this study is to see if adding a numbing medicine, xylocaine, to the nasal midazolam makes giving the midazolam easier and more comfortable without affecting how the midazolam works as a sedative.

DETAILED DESCRIPTION:
Midazolam is often given before surgery to sedate a patient before anesthesia is given. Children are often given a small dose either by mouth or squirted into the nose. Children will often spit out the oral midazolam, making it difficult to know how much medicine, if any, they have received. Giving midazolam into the nose is more reliable, but children may complain of pain, stinging, and may become upset due to the discomfort. Nosebleeds may also occur when midazolam is squirted alone into the nose. The purpose of this study is to see if adding a numbing medicine, xylocaine, to the nasal midazolam makes giving the midazolam easier and more comfortable without affecting how the midazolam works as a sedative.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 18 months-7 years, scheduled for a minor otolaryngology (ENT) surgical procedure requiring mask anesthesia
2. American Society of Anesthesiologists (ASA) Class 1 or 2
3. Parent willing and able to provide written informed consent
4. Parent willing and able to complete the OBD VAS

Exclusion Criteria:

1. ASA Class 3 or greater
2. History of allergy to midazolam or xylocaine
3. Presence of acute respiratory infection at time of surgery
4. Parent unwilling or unable to provide informed consent
5. Parent unwilling or unable to complete the OBD VAS

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: david Ullman, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Placebo: Control patients received intranasal saline.
- Nasal Midazolam Only: Patients received 0.2 mg/kg of intranasal midazolam
- Midazolam Plus Xylocaine: Patients received 0.2 mg/kg intranasal midazolam plus xylocaine 4% in a dose based on 25% of the volume of the midazolam.
Period: Overall Study
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: It was determined that a minimum of 15 patients (5 in each group) were necessary for baseline statistical analysis of this pilot study, to be used in performing a formal power analysis and sample size calculation. However, limitations in the number of providers and eligible patients during the two-year study period prevented further recruitment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.2 (2.2) | 4.0 (1.2) | 4.0 (2.0) | 3.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 3 | 4 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
American Society of Anesthesiologists Physical Status Class [Number; unit: participants] — ASA Class 1: A healthy patient, ASA Class 2: A patient with mild systemic disease
  participants
    ASA Class 1 | 1 | 2 | 2 | 5
    ASA Class 2 | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Sedation Scale Score
Description: Measured by the administering RN. Measured as: agitated, alert, calm, drowsy, asleep.
Time Frame: 10 minutes post-sedation
Population: participants with available data at this time point
Measure: Number; unit: participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 4 | 4 | 5
participants
  Agitated | 0 | 0 | 0
  Alert | 1 | 2 | 2
  Calm | 3 | 2 | 3
  Drowsy | 0 | 0 | 0
  Asleep | 0 | 0 | 0
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.99, Chi-squared

2. Primary Outcome: Sedation Scale Score
Description: Measured by the administering RN. Measured as: agitated, alert, calm, drowsy, asleep.
Time Frame: 15 minutes post-sedation
Population: participants with available data at this time point
Measure: Number; unit: participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 4 | 3 | 3
participants
  Agitated | 0 | 0 | 0
  Alert | 1 | 1 | 1
  Calm | 3 | 2 | 2
  Drowsy | 0 | 0 | 0
  Asleep | 0 | 0 | 0
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.99, Chi-squared

3. Primary Outcome: Time From Administration to Discharge
Time Frame: Minutes from administration to discharge
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 5 | 5 | 5
minutes | 87.0 (21.9) | 74.2 (9.6) | 97.0 (18.9)
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.26, Kruskal-Wallis

4. Secondary Outcome: Parental Observed Behavioral Distress Score
Description: Measured by the accompanying parent using a Visual Analog Scale. The scale ranges from a minimum score of 0 (no distress at all) to a maximum of 10 (most distress possible).
Time Frame: 1 minute post-administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 5 | 5 | 5
units on a scale | 0.08 (0.2) | 3.10 (2.4) | 1.96 (1.5)
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.02, Kruskal-Wallis

5. Secondary Outcome: RN Observed Behavioral Distress Score
Description: Measured by the administering RN using a Visual Analog Scale. The scale ranges from a minimum score of 0 (no distress at all) to a maximum of 10 (most distress possible).
Time Frame: 1 minute post-administration
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Saline Placebo: Control patients will received intranasal saline.
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 5 | 5 | 5
units on a scale | 0.1 (0.2) | 2.4 (3.0) | 1.9 (1.7)
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.04, Kruskal-Wallis

6. Secondary Outcome: Verbal Complaint
Description: Recorded by the administering RN at the time of administration.
Time Frame: At time of administration
Measure: Number; unit: participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 5 | 5 | 5
participants
  No Complaint | 3 | 1 | 2
  Complaint Reported | 2 | 4 | 3
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.73, Chi-squared

7. Secondary Outcome: Verbal Complaints
Description: Recorded by the administering RN at one minute post-administration
Time Frame: 1 minute post-administration
Measure: Number; unit: participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 5 | 5 | 5
participants
  No Complaint | 5 | 3 | 4
  Complaint Reported | 0 | 2 | 1
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority or Other; p = 0.73, Chi-squared

ADVERSE EVENTS:
Time Frame: During hospital stay.
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Limitations in the number of providers and eligible patients during the two-year study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes